CLINICAL TRIAL: NCT05065814
Title: The Effect of Vitamin D Deficiency on Exercise Capacity and Peripheral Muscle Strength
Brief Title: Connective Tissue Diseases and Vitamin D Deficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Fulden Sarı, research assistant, Gazi University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 205
Record Dates: First submitted 2021-07-15; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Connective Tissue Diseases
Keywords: connective tissue disease; muscle strength; exercise capacity
MeSH Terms: conditions — Connective Tissue Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Systemic lupus erythematosus group (Other): Demographic information of systemic lupus erythematosus patients who accepted to participate in the study will be obtained, and respiratory and peripheral muscle strength and exercise capacity of the patients will be evaluated with a 6-minute walking test. Patients will be asked to complete the International Physical Activity Questionnaire, the numerical pain questionnaire, the Short Form-36, and the Hospital Anxiety and Depression Questionnaire. In addition, Modified Medical Research Council Dyspnea Scale will be applied by the interviewer.
  Interventions: Other: Systemic lupus erythematosus group
- Systemic sclerosis group (Other): Demographic information of systemic sclerosis who accepted to participate in the study will be obtained, and respiratory and peripheral muscle strength and exercise capacity of the patients will be evaluated with a 6-minute walking test. Patients will be asked to complete the International Physical Activity Questionnaire, the numerical pain questionnaire, the Short Form-36, and the Hospital Anxiety and Depression Questionnaire. In addition, Modified Medical Research Council Dyspnea Scale will be applied by the interviewer.
  Interventions: Other: Systemic sclerosis group
- Healthy control group (Other): Healthy individuals with no chronic diseases who agreed to participate in the study and gave their consent will be included in the study.
  Interventions: Other: Healthy control group

INTERVENTIONS:
Other: Systemic lupus erythematosus group — Demographic information of systemic lupus erythematosus who accepted to participate in the study will be obtained, and respiratory and peripheral muscle strength and exercise capacity of the patients will be evaluated with a 6-minute walking test. Patients will be asked to complete the International Physical Activity Questionnaire, the numerical pain questionnaire, the Short Form-36, and the Hospital Anxiety and Depression Questionnaire. In addition, Modified Medical Research Council Dyspnea Scale will be applied by the interviewer.
  Arms: Systemic lupus erythematosus group
Other: Systemic sclerosis group — Demographic information of Systemic sclerosis who accepted to participate in the study will be obtained, and respiratory and peripheral muscle strength and exercise capacity of the patients will be evaluated with a 6-minute walking test. Patients will be asked to complete the International Physical Activity Questionnaire, the numerical pain questionnaire, the Short Form-36, and the Hospital Anxiety and Depression Questionnaire. In addition, Modified Medical Research Council Dyspnea Scale will be applied by the interviewer.
  Arms: Systemic sclerosis group
Other: Healthy control group — Healthy individuals with no chronic diseases who agreed to participate in the study and gave their consent will be included in the study.
  Arms: Healthy control group

SUMMARY:
Connective tissue disease (CTD) covers all heterogeneous and broad immunological diseases. These immunological diseases are characterized by inflammation, tissue damage, and abnormal repair. Disorders such as fibrotic tissue or loss of function are seen in the degeneration of the target organ. There is a complex relationship between genetic and environmental factors on the basis of these disorders.

Vitamin D deficiency has been frequently observed in autoimmune diseases such as systemic lupus erythematosus, diabetes mellitus, and rheumatoid arthritis. Vitamin D deficiency is primarily seen with musculoskeletal complaints and is an early warning of osteomalacia. Muscle weakness is most common in the trunk, shoulders and hips. It is characterized by difficulty in climbing stairs, getting up from sitting or lying position, feeling of heaviness in the legs, duck-like gait, difficulty getting up from a chair, fatigue easily, inability to lift objects with arms and hands. Patients experience decreased exercise capacity as a result of pain and muscle weakness. In addition, vitamin D deficiency causes smooth muscle contraction and an increase in airway inflammation. As a result, it was observed that the disease course and symptoms were more severe in CVD patients with vitamin D deficiency. In a study conducted with rheumatoid arthritis patients, the quality of life, physical activity and depression levels of patients with vitamin D deficiency were compared with the control group. The evaluation parameters of rheumatoid arthritis patients were worse than the control group. Vitamin D levels were compared with sleep, anxiety and depression levels in patients with systemic lupus erythematosus. A positive relationship was found between vitamin D deficiency and sleep disturbance level. It has been observed that the life expectancy of patients with connective tissue disease is significantly reduced compared to healthy ones. Exercise capacity and oxygen consumption decreased in these patients.

DETAILED DESCRIPTION:
Outpatient connective tissue disease patients (systemic sclerosis and systemic lupus erythematosus) with stable medical conditions will be referred for physiotherapy and rehabilitation after being examined by the relevant physician. Physiotherapy evaluation will be made by the physiotherapist. In addition; healthy individuals who accepted and gave consent to participate in the study without any chronic disease for the healthy control group will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable general condition treated with standard medical treatment
* Patients between the ages of 18-65

Exclusion Criteria:

* Patients who cannot cooperate with the assessment
* Those who have orthopedic problems or neurological diseases that will affect the evaluation of functional capacity
* Patients with pneumonia or any acute infection at the time of assessment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Functional exercise capacity | First day
  Functional exercise capacity will be evaluated with the 6-minute walk test according to the European Respiratory Society and American Thoracic Society (ATS/ERS) criteria.
Peripheral muscle strength | First day
  Shoulder flexors, shoulder abductors, knee extensors and hip flexors of the patients will be evaluated with a portable digital hand dynamometer.

SECONDARY OUTCOMES:
Numerical Evaluation Scale-Pain | First day
  The Numeric Rating Scale (NRS) was used to determine the pain level of the patients at rest, activity and at night. Patients are asked to mark the numbers between 0 and 10 at the time of assessment, in terms of rest, activity and night pain.
Modified Medical Research Council Dyspnea Scale | First day
  Assessment of dyspnea was assessed with the Modified Medical Research Council (MMRC) dyspnea scale. The MMRC is a category scale consisting of 5 statements about dyspnea, scored between 0-4.
Hospital Anxiety and Depression Scale | First day
  A valid and reliable Turkish Hospital Anxiety and Depression Scale (HADS) was used to determine the anxiety and depression levels of the patients. In the questionnaire consisting of a total of 14 questions, odd-numbered questions assess anxiety and even-numbered questions assess depression. It has two subgroups, anxiety (HADS-A) and depression (HADS-D). The lowest score that patients can get from both subgroups is 0, and the highest score is 21.
Fatigue Severity Scale | First day
  It will be evaluated with the Fatigue Severity Scale (FSS). It is a scale used by the individual to determine the perception of fatigue. The scale consists of nine items, each item is scored between 1-7. An increase in the total score obtained from the scale indicates that the severity of fatigue of the individual increases.
International Physical Activity Questionnaire-short form | First day
  Physical activity level was evaluated with Turkish valid and reliable International Physical Activity (IPAQ) questionnaire. The questionnaire consisting of 7 questions gives information about the time spent in walking, moderate-to-vigorous and vigorous activities. The time spent sitting is considered as a separate question. A score is obtained in total score metabolic equivalent (MET)-minutes. According to the result, physical activity level is classified as 'inactive', 'minimally active' and 'very active'.
Short-form 36 | First day
  Quality of life will be evaluated with the Short-form 36 (SF-36), which is completed considering the last 4 weeks. SF-36 questionnaire; It includes a total of 36 questions in eight subgroups: physical function, physical role difficulty, pain, general health, vitality, social function, emotional role difficulty and mental health. Separate scores are calculated for eight subgroups. SF-36 evaluates the negative and positive aspects of the general health condition together. Subgroup scores range from 0 to 100, with a high score indicating good health.

CONTACTS AND LOCATIONS:
Overall Officials: Deran OSKAY, Prof, Study Director — Gazi University
Locations (1):
- Gazi University, Çankaya, Ankara, Turkey (Türkiye)